CLINICAL TRIAL: NCT00005890
Title: Diagnostic Study of Adrenal Cortical Function in Children With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Purpose: Diagnostic
Other Study IDs: NCRR-M01RR08084-0043; CHMC-C-96-3-5
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Septic Shock
Keywords: immunologic disorders and infectious disorders; rare disease; sepsis; septic shock
MeSH Terms: conditions — Shock, Septic; Immune System Diseases; Communicable Diseases; Rare Diseases; Sepsis | interventions — Adrenocorticotropic Hormone

INTERVENTIONS:
Drug: corticotropin

SUMMARY:
OBJECTIVES:

I. Examine adrenal cortical function and the incidence of adrenal dysfunction in children with septic shock.

II. Examine the mortality, length of stay in the PICU, and incidence of multiorgan failure in children with adrenal dysfunction and septic shock.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo a corticotropin stimulation test within 8 hours of admission to the PICU. Blood samples for plasma cortisol and corticotropin levels are drawn at time 0 followed by corticotropin 1-24 IV. Additional cortisol levels are drawn at 30 and 60 minutes. Corticotropin is measured by immunoradiometric assay and cortisol is measured by radioimmunoassay. Mean arterial blood pressure, heart rate, and respiratory rate are recorded at baseline and at 60 minutes.

Patients receive routine management for septic shock and multiple organ system failure.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Patients admitted to the PICU with septic shock; Hypotension (systolic blood pressure less than 2 standard deviations below age normal) plus 3 or more of the following: temperature greater than 38 or less than 36 degrees Celsius; heart rate greater than 90th percentile for age; respiratory rate greater than 90th percentile for age; WBC greater than 12,000/mm3 or less than 4,000/mm3 or greater than 10% band forms; perfusion abnormalities including lactic acidosis, oliguria, or an acute alteration in mental status

Arterial or central venous catheter in place

--Prior/Concurrent Therapy--

At least one month since prior corticosteroids

--Patient Characteristics--

Renal: No nephrotic syndrome requiring glucocorticoids

Pulmonary: No asthma requiring glucocorticoids

Other: No condition requiring glucocorticoids (e.g., adrenal insufficiency); No uncontrolled diabetes mellitus; No prior adrenal dysfunction (plasma cortisol concentration less than 19 mcg/dL 30 and 60 minutes post corticotropin stimulation); No hypersensitivity to corticotropin

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56
Dates: Start 1996-03

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Brilli, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio, United States